CLINICAL TRIAL: NCT03313323
Title: Uptake and Biodistribution of 89Zirconium-labeled Ipilimumab in Ipilimumab Treated Patients With Metastatic Melanoma
Acronym: Zirconipi
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, A.J.M. van den Eertwegh, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015.300
Record Dates: First submitted 2017-08-08; First posted 2017-10-18 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Melanoma
Keywords: Immuno-PET; Ipilimumab; Immunotherapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Zirconium-ipilimumab (Experimental): Zirconium-ipilimumab is an experimental tracer and is administered at start of ipilimumab treatment and after second infusion 3 weeks later
  Interventions: Biological: 89Zirconium-labeled ipilimumab

INTERVENTIONS:
Biological: 89Zirconium-labeled ipilimumab — Metastatic melanoma patients, who are treated with ipilimumab (3 mg/kg), will be infused with 89Zr-labeled ipilimumab within 2 hours after injection of the first and second standard ipilimumab doses. Peripheral blood mononuclear cells (PBMCs) will be collected for immunomonitoring.

SUMMARY:
Rationale:

Ipilimumab, a monoclonal antibody targeting CTLA-4, is approved for the treatment of metastatic melanoma and significantly increases median overall survival. However, use of this drug is associated with immune related adverse events (IRAEs) like colitis, hepatitis, dermatitis, alveolitis and hypophysitis in 10-40% of the patients. In general IRAEs are manageable by cessation of ipilimumab in combination with treatment with corticosteroids or TNF-alpha blockade but they can be severe or even life-threatening. In addition, treatment with ipilimumab is expensive. Because of the high costs and the potential serious toxicity of ipilimumab, it is of great importance to identify biomarkers that correlate with clinical activity and can be used to select patients that will benefit from CTLA-4 blockade therapy.

The investigators hypothesize that differences in response to treatment with ipilimumab are due to variability in the pharmacodynamics and -kinetics of the antibody. It is hypothesized that patients who do not respond to treatment with ipilimumab have lower drug levels in tumor tissues as compared to patients with a good response to therapy. In addition, the investigators hypothesize that IRAEs are associated with high drug levels in the affected tissue.

To visualize molecular interactions a novel technique is used in which positron emission tomography (PET) is combined with labeled monoclonal antibodies. Because ipilimumab induces activation of T-lymphocytes it is hypothesized that uptake of 89Zr-ipilimumab in tumor lesions and normal tissue is different (i.e. higher) after the second administration of ipilimumab (3 weeks after first injection). Therefore immuno-PET scans will be performed after the first and after the second injection of ipilimumab.

Objective:

Part one: The primary objective is:

1. To assess uptake (visual and quantitative) of 89Zr-ipilimumab in tumor lesions and biodistribution at two timepoints (at start of ipilimumab therapy and after the second injection 3 weeks later).

The secondary objectives are:

1. To determine the correlation between tumor targeting of ipilimumab and response to therapy.
2. To assess uptake (visual and quantitative) of 89Zr-ipilimumab in normal tissues.
3. To determine de correlation between organ targeting and toxicity

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Advanced/metastatic melanoma.
* Scheduled for treatment with ipilimumab.
* Age ≥ 18 years.
* Histological or cytological documentation of cancer is required.
* WHO Performance Status of 0 or 1.
* At least 1 measurable lesion.
* Signed informed consent must be obtained prior to any study procedures.
* Patients must be able to adhere to the study appointments and other protocol requirements.

Exclusion Criteria:

* Previous exposure to ipilimumab.
* Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start treatment. Both men and women enrolled in this trial must agree to use adequate barrier birth control measures (e.g. cervical cap, condom and diaphragm) during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between study drug and oral contraceptives. Concomitant use of oral and barrier contraceptives is advised. Contraception is necessary for at least 6 months after receiving study drug.
* Concurrent anticancer chemotherapy, immunotherapy or investigational drug therapy during the study or within 4 weeks after starting the study drug.
* Radiotherapy of target lesions during study or within 4 weeks after starting the study drug. Palliative radiotherapy will be allowed.
* Major surgery within 28 days of start of study drug.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
The detection of 89Zr-ipilimumab in tumor lesions | 3 weeks
  The detection (visual and quantitative) of 89Zr-ipilimumab in tumor lesions (the short axis diameter of a measurable tumor lesion is ≥1 cm. The five largest lesions will be used for evaluation).

SECONDARY OUTCOMES:
The visual detection of 89Zr-ipilimumab in normal tissue | 3 weeks
  The visual detection of 89Zr-ipilimumab in normal tissue after the first injection of ipilimumab and after the second injection 3 weeks later. Visual: Description of the biodistribution.
The quantitative detection of 89Zr-ipilimumab in normal tissue | 3 weeks
  The quantitative detection of 89Zr-ipilimumab in normal tissue after the first injection of ipilimumab and after the second injection 3 weeks later. Quantitative: The % uptake (of total injected) 89Zr-ipilimumab in normal tissue, measured in VOI's.
Comparison between uptake of 89Zr-ipilimumab | 3 weeks
  Comparison between uptake (SUVmean and SUVpeak) of 89Zr-ipilimumab after the first injection of ipilimumab and after the second injection 3 weeks later.
Clinical outcome (response) | Every 12 weeks, from date of starting therapy until the date of first documented progression or date of death from any cause, whichever came first. Assessed through study completion, an average of 1 year
  Response after starting therapy with ipilimumab at 12 and 24 weeks and every 12 weeks thereafter
Clinical outcome (survival) | Through study completion, an average of 1 year
  Overall survival
Side effects | Until 30 days after the last immuno-PET scan
  * Adverse events using Common Terminology Criteria Adverse Events, version 4.0 (CTCAE 4.0)
  * Correlation between side effects of ipilimumab and uptake of 89Zr-ipilimumab in normal tissue
Pharmacokinetics of 89Zr-ipilimumab | 144 hours after first injection of 89Zr-ipilimumab
  Pharmacokinetics of 89Zr-ipilimumab. The concentration of ipilimumab in blood samples will be measured at t = 5, 30, 60, 120 minutes and 72, 144 hours after injection of 89Zr-ipilimumab in the first three patients.
CTLA-4+CD4+ expression of PBMCs | Before start of ipilimumab and during treatment, up to 11 weeks
Immunohistochemical analysis | 3 weeks
  Immunohistochemical analysis (% of tissue with inflammatory infiltrate and characterization of intratumoral T-lymphocytes (CD4, CD8, HLA-DR, FOX-P3, CTLA-4) of tumor biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Alfonsus JM van den Eertwegh, Prof.dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No